CLINICAL TRIAL: NCT06718556
Title: Virtual Reality Intervention for Visual Perception in Schizophrenia-A Single Blind Pilot Randomized Controlled Trial
Brief Title: Virtual Reality for Visual Perception on Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Assoc Prof, Vice Dean, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/08-07
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Schizophenia Disorder; Virtual Reality; Visual Perception
Keywords: schizophrenia; virtual reality; visual perception; client centered; intervention
MeSH Terms: conditions — Schizophrenia | interventions — Person-Centered Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality group (Experimental): The intervention procedure was planned to consist of 8 weeks, 3 days a week and 45-minute sessions in total.
  In this intervention group, a virtual reality intervention was applied in addition to the client-centered intervention applied to both groups.
  Interventions: Behavioral: Virtual reality; Behavioral: Client-centered
- Control group (Experimental): Client-centered intervention procedure was applied to the control group. The intervention procedure was planned to consist of 8 weeks, 3 days a week and 45-minute sessions in total.
  Interventions: Behavioral: Client-centered

INTERVENTIONS:
Behavioral: Virtual reality — The virtual reality intervention program was carried out in a 30-meter2 area covered with soft ground to prevent injuries. "The Microsoft Kinect for Xbox 360" was used for the virtual reality intervention. For the current study, a team of experts was formed to select the games to be used within the virtual reality intervention program. This team determined which skills were required for the games to be run successfully, which skills could be developed, which games were purposeful, and independently observed each game. As a result, 9 different games were chosen. Since all games involve similarly intense visual, cognitive and motor skill requirements, game selection was left to the participants' preference during the intervention process to encourage motivation and participation. The virtual reality intervention procedure was created by utilizing the literature
  Arms: Virtual reality group
Behavioral: Client-centered — The client-centered (CC) intervention procedure for individuals with schizophrenia was created using literature and the intervention procedure is presented below:
  1. Active Communication and Evaluation
  2. Daily Routine, Roles, and Occupational Performance
  3. Strengths and Barriers
  4. Intervention Program Development
  5. Implementation of the intervention program
  6. Feedback and Revision:

SUMMARY:
Researchers have stated in the literature that visual perception is negatively affected in schizophrenia. In recent years, virtual reality interventions have become popular in the treatment of schizophrenia. However, there are no virtual reality studies that directly focus on visual perception. This study was planned to examine the effect of virtual reality intervention on visual perception in individuals with schizophrenia.

DETAILED DESCRIPTION:
The current study was planned as a pilot randomized controlled study and the study was conducted using the CONSORT checklist. Participants who met the inclusion and exclusion criteria and signed the written consent form were divided into 2 groups by simple random method. VR and client-centered intervention procedure was applied to the intervention group, and client-centered intervention procedure was applied to the control group. The intervention procedure was planned to consist of 8 weeks, 3 days a week and 45-minute sessions in total.

The study evaluated 64 individuals diagnosed with schizophrenia. 57 individuals with schizophrenia who completed the assessment and met the inclusion/exclusion criteria were included. These 57 individuals were given a number on the computer and then randomization was performed on the computer, and 29 participants were included in the VR group and 28 in the control group. During the intervention process, two individuals in each group who could not participate regularly were excluded from the study and the study was completed with 53 participants. The randomization process was carried out by a researcher who was independent of the study and did not know the assessment and intervention process.

Measurement Sociodemographic information of the participants, such as age, gender, marital status, education and employment status, was collected. After the sociodemographic data were collected, the Motor-Free Visual Perception Test-3rd Edition (MVPT-3) was used to evaluate the visual perceptions of the participants before and after the interventions.

Interventions Virtual reality intervention procedure The VR intervention program was carried out in a 30-meter2 area covered with soft ground to prevent injuries. "The Microsoft Kinect for Xbox 360" was used for the VR intervention. For the current study, a team of experts was formed to select the games to be used within the VR intervention program. This team determined which skills were required for the games to be run successfully, which skills could be developed, which games were purposeful, and independently observed each game. As a result, 9 different games were chosen. The VR intervention procedure was created by utilizing the literature.

Client-centered intervention procedure

The client-centered (CC) intervention procedure for individuals with schizophrenia was created using literature. This intervention procedure consists of 6 steps. These steps are:

1. Active Communication and Evaluation
2. Daily Routine, Roles, and Occupational Performance
3. Strengths and Barriers
4. Intervention Program Development
5. Implementation of the intervention program
6. Feedback and Revision In addition, studies have been conducted on both visual perception and social skills with personalized targeted tasks. In order to develop visual perception, interventions were made to the participants to develop the parameters of visual perception skills such as visual memory, visual closure, shape-ground perception, visual discrimination, visual completion, spatial orientation, etc., which are sub-parameters of visual perception skills. In addition, studies have been conducted to develop social skills, especially basic social skills such as "listening to others, making requests, expressing positive emotions and expressing unpleasant emotions".

Statistically analysis Data were analyzed with SPSS version 29.0 statistical software package program. The normality of the data was analyzed by using Kolmogorov-Smirnov test. Nonparametric tests were used because the data did not show a normal distribution. Differences between groups were analyzed with chi-square test for nominal data. Comparisons between the groups were conducted by using the Mann-Whitney U test. Pre- to post-intervention changes within the groups were analyzed with the Wilcoxon signed-rank test. Significance was evaluated at levels of 0.05. Effect size was calculated by using the means and standard deviations of the groups. Effect size benchmarks were determined as <0.30, 0.30-0.80, and >0.80 and considered small, moderate, and strong, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia by a psychiatrist according to DSM-5 criteria.
* Age between t 18 and 65.
* Ability to understand and follow verbal instructions.
* Active and voluntary participation in the study.
* Being stated to be in clinical remission by a psychiatrist.

Exclusion Criteria:

* Having any chronic disease (neurological, orthopedic, psychiatric, cancer, epilepsy etc.) in addition to schizophrenia that may affect the study.
* Presence of mental retardation.
* Inability to complete the intervention procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Motor-Free Visual Perception Test-3rd Edition-MVPT 3 | 30 minutes
  MVPT-3 is a widely used scale for the assessment of visual perception. The test consists of nine main subheadings, namely visual discrimination (1-8), shape formation (9-13), visual memory-I (14-21), visual closure-I (22-34), visual discrimination (35-45), spatial orientation (46-50), figure-ground (51-55), visual closure-II (56-60) and visual memory-II (61-65), and consists of 65 items. This test is administered individually to participants between the ages of four and ninety-five. The first 40 items are administered to children between the ages of four and ten, and the remaining 51 items from item 14 to item 65 are for individuals aged ten and over. In the study conducted by Metin and Aral for Turkish validity, the Cronbach's alpha coefficient of the test was determined as 0.85.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No